CLINICAL TRIAL: NCT02593266
Title: A Pilot Randomized Controlled Trial of a Preventive Intervention Program for Chilean Families With Depressed Parents
Brief Title: A Trial of a Preventive Intervention Program for Chilean Families With Depressed Parents
Acronym: FamilyTalkCL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Boston Children's Hospital (Other); Wellesley College (Other)
Responsible Party: Principal Investigator, Matias Irarrazaval, Dr. Matias Irarrazaval MD MPH, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FONDECYT-11130615
Record Dates: First submitted 2015-05-28; First posted 2015-11-02 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Depression
Keywords: Prevention; Family; Intervention; Depression; Children
MeSH Terms: conditions — Depression | interventions — PIP protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): weekly sessions of PIP for depression.
  Interventions: Behavioral: Preventive Intervention Program (PIP) for depression
- Waiting list control group (No Intervention): This is treatment as usual.

INTERVENTIONS:
Behavioral: Preventive Intervention Program (PIP) for depression — Manualized intervention designed by Beardslee and colleagues (Beardslee et al., 2003) It is a program based on cognitive behavioural therapy, narrative therapy and systemic therapy. It is divided in 7 modules which are imparted weekly in the family home by 2 'preventionists' (therapists trained to deliver the intervention)
  * Module 1: Depression and family
  * Module 2: Psychoeducation about depression
  * Module 3:The child's perspective on their parent's depression
  * Module 4: Skills development
  * Module 5: Preparation for the family session
  * Module 6: Family session
  * Module 7: Revision and future planning
  * Follow-up
  Arms: Intervention Group

SUMMARY:
The overall aim of this pilot study is to evaluate the acceptability and feasibility of an adaptation of Beardslee's 'Preventive Intervention Program (PIP) for Depression' in Chilean families.

The PIP is a family intervention directed towards strengthening family functioning and enhancing resilience in children of depressed parents. It comprises several modules that work on psycho-education and skill development within the family nucleus.

A single-blind randomized controlled trial will be conducted with two arms, the intervention arm (n=32) which will receive a home-based PIP for depression, and the TAU arm (n=32).

DETAILED DESCRIPTION:
Being a child with depressed parents is associated with poor health and academic outcomes as well as having four times the likelihood of developing a mood disorder compared to children of non-depressed parents.

Objectives: To evaluate acceptability and feasibility of an adaptation of Beardslee's 'Preventive Intervention Program (PIP) for Depression' in Chilean families, and to measure the clinical effects of this intervention.

Participants: Parents with an episode of Depression in the past 3 months with at least one non-depressed child between the ages of 6-12.

Design: single-blind randomized controlled trial with two groups; the intervention group (n=32), which will receive a home-based PIP for depression, and the treatment-as-usual control group (n=32).

Results: Acceptability and feasibility will be measured by determining whether the trial was successfully conducted and well received by the families and preventionists. Recruitment and delivery of the intervention will be assessed as well as whether there was appropriate response and follow-up, and whether the objectives of the study were reached. Secondary outcomes will look at depressive symptoms, family function, psycho-education, parental competence, adaptive behavior and resilience in children.

Follow-up times: T = 0 baseline, T= 2 months (post-intervention), T=5 months, T=8 months, T=11 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are currently undergoing a depressive episode or have done so in the past 3 months.

Exclusion Criteria:

For parents:

* Alcohol or drug dependence or abuse as assessed by the MINI or being in treatment for substance use.
* Psychosis, personality disorder, bipolar disorder or suicide ideation as assessed by the MINI.
* Having a relationship crisis with current partner. Assessed by self-report or by having attended couple's therapy in the past month.
* Attending family therapy.

For children:

* Being outside the age range of 6-12 years at the time of recruitment.
* Intellectual disability
* Having depression as assessed by the MINI Kid
* Being in treatment for a psychiatric disorder or having taken psychotropic medication in the last month.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
acceptability | 7 weeks
  The acceptability of the intervention will be evaluated through qualitative questionnaires.
feasibility | 7 weeks
  Feasibility will be assessed by looking at the number of families succesfully completing the study.

SECONDARY OUTCOMES:
Depressive symptoms in children | 11 months
  scores on the depression scale CDI
Depressive symptoms in parents | 11 months
  scores on the depression scale BDI
Family functioning | 11 months
  scores on the FACES-II scale
Parental competence | 11 months
  scores on the E2P scale
Adaptive behaviour in children | 11 months
  scores on the CBCL scale
resilience in children | 11 months
  scores on the ERE scale

CONTACTS AND LOCATIONS:
Overall Officials: Matias Irarrazaval, PhD, Principal Investigator — University of Chile
Locations (1):
- Clinica psiquiatrica Universitaria, Santiago, Chile

REFERENCES:
- [Derived] de Angel V, Prieto F, Gladstone TR, Beardslee WR, Irarrazaval M. The feasibility and acceptability of a preventive intervention programme for children with depressed parents: study protocol for a randomised controlled trial. Trials. 2016 May 6;17(1):237. doi: 10.1186/s13063-016-1348-7. PMID 27153835
- See also: Collaborator's website — http://www.fampod.org